CLINICAL TRIAL: NCT01100931
Title: A Phase I/II Study of Paclitaxel, Carboplatin and YM155 (Survivin Suppressor) in Subjects With Solid Tumors (Phase I) and Advanced Non-Small Cell Lung Carcinoma (Phase II)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100051; 10-C-0051
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: NSCLC; Solid Tumors
Keywords: NSCLC; Solid Tumors; YM155; Survivin; Non Small-Cell Lung Cancer; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sepantronium; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM155 in Solid Tumors (Experimental): Phase I: Doses were given at different dose levels until the maximum tolerated dose (MTD) was reached. Dose level 1: 3.6 mg/m^2, dose level 2:5 mg/m^2 , dose level 3:6 mg/m^2, dose level 4:8 mg/m^2, dose level 5:10 mg/m^2 (MTD), dose level 6:12 mg/m^2. Doses were given by continuous intravenous infusion over 72 hours every 21 days.Three patients were enrolled at each dose level in the absence of dose limiting toxicity (DLT). A DLT is defined as adverse events occurring during the first cycle of therapy (e.g. every 21 days).
  Phase II: 10 mg/m^2 (MTD)intravenous infusion over 72 hours every 21 days.
  Interventions: Drug: YM155; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: YM155 — Phase I: Doses were given at different dose levels until the maximum tolerated dose (MTD) was reached. Dose level 1: 3.6 mg/m^2, dose level 2:5 mg/m^2 , dose level 3:6 mg/m^2, dose level 4:8 mg/m^2, dose level 5:10 mg/m^2 (MTD), dose level 6:12 mg/m^2. Doses were given by continuous intravenous infusion over 72 hours every 21 days.Three patients were enrolled at each dose level in the absence of dose limiting toxicity (DLT). A DLT is defined as adverse events occurring during the first cycle of therapy (e.g. every 21 days).
  Phase II: 10 mg/m^2 (MTD)intravenous infusion over 72 hours every 21 days.
Drug: Carboplatin — Area under curve (AUC) of 6 intravenous on day 1
  Other Names: Paraplatin
Drug: Paclitaxel — 200 mg/m^2 intravenous on day 1
  Other Names: Taxol

SUMMARY:
Background:

* Carboplatin-paclitaxel is a commonly used chemotherapy combination for advanced non-small-cell lung carcinoma (NSCLC) and other solid tumors. In a randomized clinical trial, the combination of carboplatin, paclitaxel, and the additional chemotherapy drug bevacizumab had a better response rate and survival compared to carboplatin and paclitaxel alone. However, this trial treated only patients with a specific diagnosis and treatment risks. Further research is needed to determine whether this combination is useful for other diagnoses.
* YM155 is a drug that targets a type of chemical often found in cancer cells. It has been investigated in several phase I and phase II clinical trials, and it has been shown to be well tolerated and moderately effective in treating advanced NSCLC in patients who had not responded well to one or two standard treatments.

Objectives:

- To determine the efficacy of the combination of carboplatin, paclitaxel, and YM155 in the treatment of non-small-cell lung cancer.

Eligibility:

- Individuals 18 years of age and older who have been diagnosed with advanced non-small-cell lung carcinoma or other solid tumors for which standard therapy is not likely to be effective.

Design:

* Before the start of the study, participants will be screened with a medical history, blood tests, imaging scans of the affected areas, tumor biopsies, and other tests as directed by the study doctors.
* Participants will be treated for six 21-day cycles, or 18 weeks of treatment. Each cycle will include blood tests and imaging studies as required.
* On day 1 of each cycle, participants will receive an infusion of paclitaxel and carboplatin, followed by a 4-day infusion of YM155 (through a portable electronic infusion pump).
* Participants will have a computed tomography scan or other imaging every other cycle (approximately every 6 weeks) to determine whether the therapy is affecting the cancer site.
* After the sixth cycle, participants will return for follow-up visits at least every 3 months, and will be asked to remain in contact with the researchers to allow further study of the long-term effects of the treatment.

DETAILED DESCRIPTION:
Background:

* Treatment with platinum-based doublet chemotherapy results in a median survival of 7 to 10 months in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC).
* Carboplatin-paclitaxel is a commonly used regimen in advanced NSCLC and other solid tumors. In a randomized clinical trial carboplatin, paclitaxel plus bevacizumab resulted in improved efficacy (response rate and survival) compared to carboplatin and paclitaxel alone but only patients with non-squamous histology and who were considered low risk of bleeding were treated. Improvement of survival was not confirmed in another randomized study with a different chemotherapy backbone.
* Novel treatment strategies need to be developed for advanced NSCLC.
* YM155 is a transcriptional inhibitor of survivin, an inhibitor of apoptosis protein. Pre-clinical activity of YM155 has been observed in several solid tumors, including NSCLC models and synergy was observed in combination with chemotherapeutic drugs, including carboplatin and paclitaxel.
* YM155 has been investigated in several phase I and phase II clinical trials and it has been shown to be well tolerated with the most common toxicities reported as being reversible and of grades 1 -2 in severity. In addition, as a monotherapy YM155 alone has shown modest antitumor activity in a phase II trial in advanced NSCLC in patients who had failed one or two prior chemotherapy lines.

Primary Objectives:

* In the Phase I portion of the study the primary objective will be to determine a safe and tolerable phase II dose of YM155 based upon dose limiting toxicities (DLTs) when YM155 is administered over 72 hours by continuous intravenous infusion (CIVI) every 3 weeks in combination with paclitaxel and carboplatin.
* In the Phase II portion of the study the primary objective will be to determine the objective response rate (ORR = partial response (PR)+ complete response (CR)) of YM155 in combination with carboplatin and paclitaxel in the first line treatment of patients with advanced NSCLC.

Secondary Objectives:

* In the Phase I portion of the study the secondary objective will be to determine the preliminary activity of the combination regimen based upon response rate as measured by response evaluation criteria in solid tumors [RECIST].
* In the Phase II portion of the study the secondary objectives will be to determine the median progression free survival (PFS), median overall survival (OS) and safety and tolerability of this combination regimen in this patient population.
* To assess expression of particular genes on the pretreatment tumor and pre/post treatment serum samples to evaluate the treatment effects and correlate them with clinical outcome.

Eligibility:

Phase I

- The phase I portion of the trial will be open to all patients with recurrent or advanced cancer (NSCLC and other solid tumors) for whom standard therapy offers no curative potential and also in patients for whom the carboplatin / paclitaxel regimen is considered standard of care. Patients should have received no more than one previous chemotherapy regimen.

Phase II

* Pathologically confirmed stage IIIB (malignant pleural effusion) or intravenous (IV) or recurrent NSCLC.
* No previous chemotherapy for advanced lung cancer.
* Adequate organ and bone marrow function.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Design:

* Open label phase I/II trial
* Following a Simon two-stage optimal design

ELIGIBILITY:
* INCLUSION CRITERIA:

Response should be YES

Phase 1 and 2:

1. Has a signed consent/assent been obtained by the patient or parent/legal guardian?
2. Is a male or female greater than or equal to 18 years old?
3. If patient has brain metastases, is it asymptomatic and does not require steroids or antiepileptic mediations?
4. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Karnofsky > 60%)?
5. Has adequate bone marrow, renal, and hepatic function:

   1. Absolute neutrophil count (ANC) greater than or equal to 1,500/m^3?
   2. Hemoglobin greater than or equal to 10.0g/dl?
   3. Platelets greater than or equal to 100,000/m^3?
   4. Has adequate renal function defined as serum creatinine < upper limit of normal (ULN) or calculated creatinine clearance > 60 mL/min?
   5. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times ULN?
   6. Total bilirubin less than or equal to 1.5 times ULN (in patients with evidence of Gilberts disease, elevated bilirubin should not be related to tumor or other liver diseases and should be less than or equal 2 times upper limit of normal)?
6. Has negative human immunodeficiency virus (HIV) test?
7. If female, has negative pregnancy test?
8. Both male and female patients are willing to consent to using effective contraception (hormonal, barrier method or abstinence) prior to study entry, while on treatment and at least 3 months thereafter?

Phase 1 only:

1. Has recurrent or advanced cancer for whom standard therapy offers no curative potential and also for patients for whom the carboplatin/paclitaxel regimen is considered standard of care?
2. Has received no more than one previous chemotherapy regimen?
3. Has evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria?

Phase 2 only:

1. Has histological or cytological evidence of non small cell lung cancer?
2. Has evidence of metastatic disease or stage IIIB non small cell lung cancer (NSCL) with pleural effusion is required?
3. Has no prior chemotherapy for advanced lung cancer?

   Note: Patients who received adjuvant or neo-adjuvant chemotherapy more than 12 months prior will be eligible?
4. Has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan?

EXCLUSION CRITERIA:

Response should be NO

1. Has any of the following within 6 months prior to study enrollment: myocardial infarction, unstable angina pectoris or uncontrolled angina pectoris, uncontrolled hypertension that is not controllable with antihypertensives, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, clinically significant peripheral vascular disease (Grade II or greater).
2. Has history of stroke or transient ischemic attack within 6 months?
3. Has history of pulmonary embolism, deep venous thrombosis or other thrombo-embolic event within 6 months?
4. Has psychiatric or neurologic illness that would limit compliance with study requirements?
5. Has severe active infection within 14 days requiring use of intravenous antibiotics before beginning treatment?
6. Has received any other investigational agents within 30 days of the start of treatment?
7. Has history of an active malignancy unless curatively treated and risk of recurrence of < 5% at five years, with the exception of:

   1. Adequately treated in situ carcinoma of the cervix
   2. Non-melanomatous skin cancers (basal or squamous cell)?
8. Has history of severe hypersensitivity reaction to compounds of similar chemical or biologic composition to carboplatin, paclitaxel, or medicines of similar composition to YM155?
9. Has history of a major surgical procedure, open biopsy, or a significant traumatic injury within 14 days prior to commencing treatment, or the anticipation of the need for a major surgical procedure during the course of the study?
10. Has other serious illness, medical condition or significant laboratory abnormality that may cause undue risk for the subject's safety, inhibit protocol participation, or interference with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study?
11. Phase 2 only: Has mixed tumor of any histology including small cell lung cancer?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Derived] Kelly RJ, Thomas A, Rajan A, Chun G, Lopez-Chavez A, Szabo E, Spencer S, Carter CA, Guha U, Khozin S, Poondru S, Van Sant C, Keating A, Steinberg SM, Figg W, Giaccone G. A phase I/II study of sepantronium bromide (YM155, survivin suppressor) with paclitaxel and carboplatin in patients with advanced non-small-cell lung cancer. Ann Oncol. 2013 Oct;24(10):2601-2606. doi: 10.1093/annonc/mdt249. Epub 2013 Jul 14. PMID 23857959
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0051.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient withdrew consent before starting treatment.
Groups:
- Phase I: Phase I: Doses were given at different dose levels until the maximum tolerated dose (MTD) was reached. Dose level 1: 3.6 mg/m^2, dose level 2:5 mg/m^2 , dose level 3:6 mg/m^2, dose level 4:8 mg/m^2, dose level 5:10 mg/m^2 (MTD), dose level 6:12 mg/m^2. Doses were given by continuous intravenous infusion over 72 hours every 21 days.Three patients were enrolled at each dose level in the absence of dose limiting toxicity (DLT). A DLT is defined as adverse events occurring during the first cycle of therapy (e.g. every 21 days).
- Phase II: Phase II: 10 mg/m^2 (MTD)intravenous infusion over 72 hours every 21 days.
Period: Phase I
Arm/Group | Phase I | Phase II
Started | 22 | 0
Completed | 22 | 0
Not Completed | 0 | 0
Period: Phase II
Arm/Group | Phase I | Phase II
Started | 0 | 19
Completed | 0 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.72) | 59.8 (9.51) | 61.6 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Safe and Tolerable Phase 2 Dose.
Description: Phase I: Doses were given at different dose levels until the maximum tolerated dose (MTD) was reached. Dose level 1: 3.6 mg/m^2, dose level 2:5 mg/m^2 , dose level 3:6 mg/m^2, dose level 4:8 mg/m^2, dose level 5:10 mg/m^2 (MTD), dose level 6:12 mg/m^2. Doses were given by continuous intravenous infusion over 72 hours every 21 days.Three patients were enrolled at each dose level in the absence of dose limiting toxicity (DLT). A DLT is defined as adverse events occurring during the first cycle of therapy (e.g. every 21 days).
  Phase 2 dose is based upon dose limiting toxicities experienced during cycle 1.
Time Frame: 1 year
Population: Phase I dose was variable dosing schedule to determine maximum tolerated dose (MTD) with 22 patients analyzed. Dose was variable with MTD at 10mg/m^2.
Measure: Number; unit: mg/m^2
Arm/Group | Phase I
Number analyzed (Participants) | 22
mg/m^2 | 10

2. Primary Outcome: Phase 2 Objective Response Rate (Partial Response (PR) + Complete Response (CR)).
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to 18 weeks
Population: Phase I is not included here because this outcome measure is for phase II only.
Measure: Number; unit: Participants
Arm/Group | Phase II
Number analyzed (Participants) | 19
Participants
  Complete Response | 0
  Partial Response | 2

3. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 31.5 months
Measure: Number; unit: Participants
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 22 | 19
Participants | 22 | 19

ADVERSE EVENTS:
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 10/22 | 1/19
Other Adverse Events (participants affected / at risk) | 22/22 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=22) | Phase II (N=19)
Death NOS (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=22) | Phase II (N=19)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 7 (11) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (20) | 0 (0)
Alkaline phosphatase increased (Investigations) | 5 (12) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14) | 16 (16)
Anemia (Blood and lymphatic system disorders) | 16 (61) | 7 (14)
Anorexia (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 6 (15) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Creatinine increased (Investigations) | 7 (11) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (4) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 3 (5) | 2 (2)
Electrocardiogram QT corrected interval prolong (Investigations) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye infection (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (13) | 11 (12)
Fever (General disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flu like symptoms (General disorders) | 2 (4) | 4 (4)
Flushing (Vascular disorders) | 2 (2) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 7 (7)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (8) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 6 (8) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (17) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (18) | 2 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 16 (56) | 11 (14)
Hyponatremia (Metabolism and nutrition disorders) | 12 (31) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (33) | 3 (7)
Hypotension (Vascular disorders) | 4 (4) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 5 (5)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 4 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 20 (108) | 14 (47)
lymphocyte count increased (Investigations) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 3 (3) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 1 (2) | 6 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 20 (49) | 13 (29)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (4) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (16) | 17 (23)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 12 (37) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 2 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (8)
Weight gain (Investigations) | 2 (3) | 1 (1)
Weight loss (Investigations) | 3 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
White blood cell decreased (Investigations) | 20 (74) | 12 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No